CLINICAL TRIAL: NCT07066423
Title: Impact Of Artificial Intelligence-Based Prediction of Facial Changes in Bimaxillary Protrusion Cases on Patient Motivation and Satisfaction
Brief Title: Effect of an AI Prediction Model of Facial Changes After Orthodontic Treatment of Patients With Bimaxillary Protrusion
Acronym: Ai
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Kholoud Mandour, PHD candidate, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PHD Candidate Kholoud Mandour
Record Dates: First submitted 2025-06-02; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Bimaxillary Protrusion
Keywords: Bimaxillary protrusion; prediction; Artificial intelligence; retraction; facial
MeSH Terms: conditions — Facies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ai prediction group (Experimental): The participant group that will be exposed to prediction photos and measure their motivation for the four 1st premolars extraction decision, also undergoes the orthodontic treatment.
  Interventions: Other: Ai prediction photo of the patients; Procedure: Fixed orthodontic brackets with premolars extraction
- Control group (Active Comparator): Subjects in this group will receive orthodontic treatment and answer a questionnaire about their motivation and satisfaction with the treatment, but they will not be exposed to AI prediction photos.
  Interventions: Procedure: Fixed orthodontic brackets with premolars extraction

INTERVENTIONS:
Other: Ai prediction photo of the patients — Ai prediction photo generated by specially designed ai model to help patients see how they will look after orthodontic extraction and retraction
  Arms: Ai prediction group
Procedure: Fixed orthodontic brackets with premolars extraction — Subjects will undergo orthodontic fixed brackets treatment, four premolar extractions from the mandibular and maxillary arches, followed by anterior segment retraction. This treatment will achieve dental alignment, profile, and facial enhancement.

SUMMARY:
After developing an Artificial Intelligence model to predict the facial changes of patients with bimaxillary protrusion following orthodontic extraction of premolars and tooth retraction, participants will view a prediction in the form of a picture generated by the AI model, and their motivation will be measured using a questionnaire. Their satisfaction will be evaluated using another questionnaire after they complete their treatment. A comparison will then be made between the actual results and the AI-predicted results.

DETAILED DESCRIPTION:
Subjects will be selected according to the inclusion criteria previously listed, and they will present the needed records for participating in the study. After taking initial photos of the patients before treatment, these photos will be uploaded to the AI model to generate the prediction photo, the selected subjects for the prediction group will view their AI-predicted photo, and their motivation will be evaluated by a questionnaire.

The control group will not view a prediction photo; they will answer the motivation questionnaire only.

ELIGIBILITY:
Inclusion Criteria:

1. Adult cases age range from 16 to 30 years old
2. Skeletal Bimaxillary protrusion with SNA and SNB increased
3. Dental bimaxillary protrusion with U1- SN and IMP a increased angles
4. Class I canine and molar angle classification
5. Free from any systemic disease
6. free from any dental surgery

Exclusion Criteria:

Clefts of the lip or palate and craniofacial syndromes; orthognathic patients will not be included because they do not represent the general adult orthodontic population

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Participants motivation for treatment | from three weeks to six months
  The motivation questionnaire will be performed to test if the prediction picture will affect their motivation to continue the treatment and proceed with the extraction decision. The questions will be in the multiple-choice format.
  Open-ended comments were allowed at the end of each question to collect data concerning reasons, barriers, and encouraging factors that the authors may not have considered.
  The questionnaire Arabic version will be used as it was validated by authors Felemban et al. in 2022. Based on the English version used by Chambers et al. 2019 and Laothong et al. in 2017, a modification will be added to the questionnaire regarding a question about how the prediction picture affected their motivation.
  After the treatment of each case, a 5-point Likert scale will be used to measure their satisfaction with the treatment and whether the net result matches the AI prediction, with 1 for not satisfied at all and 5 for satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Shaza Hammad, professor, Study Director — Mansoura University; Marwa Shamaa, Professor, Study Chair — Mansoura University; Ahmed Kamel, Lecturer, Study Chair — Mansoura University
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Development and accuracy of artificial intelligence-generated prediction of facial changes in orthodontic treatment: a scoping review — https://link.springer.com/article/10.1631/jzus.B2300244#citeas